CLINICAL TRIAL: NCT04586478
Title: Phase II Clinical Trial of CNCT19 Cell Injection in the Treatment of Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001205
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of CNCT19 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CNCT19.
  Interventions: Biological: single dose of CNCT19

INTERVENTIONS:
Biological: single dose of CNCT19 — Dose: 2.00 x 10^8 CNCT19 Cell Injection via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide

SUMMARY:
The study is a Phase II, single-arm, open-label, single-dose clinical trial, and its primary objective is to evaluate the efficacy and safety of CNCT19 Cell Injection in the treatment of relapsed or refractory NHL.

DETAILED DESCRIPTION:
The study is a Phase II, single-arm, open-label, single-dose clinical trial, and its primary objective is to evaluate the efficacy and safety of CNCT19 Cell Injection in the treatment of relapsed or refractory NHL. The study consists of screening period (8 weeks), treatment period (4 weeks), and follow-up period (2 years at most).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to sign the informed consent form;
2. Aged 18-75 years, male or female;
3. At screening, subjects complying with the following diagnostic and treatment requirements:

   1. Complying with CD19-positive NHL according to the WHO classification 2017, which are provided specifically as follows:

      * Diffuse large B cell lymphoma (DLBCL), not otherwise specified (NOS);
      * Primary mediastinal large B cell lymphoma (PMBCL);
      * Transformed follicular lymphoma
      * High grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high grade B cell lymphoma - not otherwise specified.
   2. Previously received≥2nd-line adequate therapy or autologous hematopoietic stem cell transplantation (ASCT), including:

      * Received at least Rituximab or other CD20 targeted drugs containing (except CD20 negative tumors) chemotherapy and
      * Received at least one chemotherapy regimen containing anthracycline;
      * Definition of line: Stable disease (SD) after receiving a first-line adequate therapy or progressive disease (PD), and SD after a second-line therapy for at least 2 cycles or PD .
   3. In relapsed or refractory status at screening:

      * Definition of relapse: Remission (including partial remission (PR) or complete remission (CR)) after treatment with at least the standard therapy regimen (it must contain Ribuximab), and then PD;
      * Definition of refractoriness:

   Non-responsiveness to the last therapy: The best response by the last therapy is SD or PD; Relapse or progression after ASCT, including: Relapse (it must be proved by biopsy) or PD within 12 months after ASCT; if a rescue therapy is received, the patient is non-responsive (SD or PD) to the last therapy;

   For transformed follicular lymphoma (TFL), patients must be treated adequately against FL, and after transformation, must have received at least once the therapy against TFL, and become relapsed or refractory after the last therapy.
4. Measurable imaging lesion at screening: Intranodal lesion must have a long diameter of more than 1.5 cm, and extranodal lesion must have a long diameter of more than 1.0 cm (per revised IWG Response Criteria 2014 in Lymphomas);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
6. Adequate bone marrow reserve, defined as:

   * Absolute neutrophil count (ANC) > 1.0×109/L;
   * Absolute lymphocyte count (ALC) ≥ 0.3×109/L;
   * Platelet (PLT) ≥50×109/L;
7. Proper organ function, complying with the following criteria (except hepatic dysfunction due to tumor cell infiltration): Aspartate aminotransferase (AST) ≤ 3 Upper Limit of Normal (ULN); Alanine aminotransferase (ALT) ≤ 3 ULN; Total serum bilirubin ≤ 2 ULN, unless there exists concurrent Gilbert syndrome; patients with Gilbert syndrome, with total serum bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN, may be included; Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula); Minimum pulmonary reserve, defined as Grade ≤ 1 dyspnea, and blood oxygen saturation > 91% at non-oxygen inhalation status; International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 ULN.
8. Vascular conditions for apheresis;
9. Women with child-bearing potential are negative in blood/urine pregnancy tests within 3 d prior to apheresis, and prior to infusion of CNCT19 cell injection infusion; any male or female patient with child-bearing potential must agree to adopt effective contraceptive measures throughout the study, and at least a year after administration of the investigational therapy. As judged by the investigator, a patient with child-bearing potential means that: He/she has normal sexual life and is biologically fertile to have children. Non-fertile female patients (i.e., complying one of the following criteria):Previously received hysterectomy, bilateral ovariectomy, or bilateral tubal ligation, or Medically confirmed ovarian failure, or Medically confirmed postmenopause (amenorrhea of at least 12 consecutive months).

Exclusion Criteria:

1. Patients with active central nervous system (CNS) lymphoma (a patient with CNS disease symptoms must receive lumbar puncture and MRI/CT to exclude CNS lymphoma).
2. Patients with existing central nervous system disease or with a history of central nervous system disease, e.g., epileptic seizure, cerebral ischemia/hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellum disease, organic brain syndrome, mental disease, or any autoimmune disease involved with central nervous system.
3. Patients receiving any of the following drugs or therapies within the specified period prior to apheresis:

   * Alemtuzumab within 6 months prior to apheresis;
   * Cladribine within 3 months prior to apheresis;
   * Anti-CD20 monoclonal antibody within 7 d prior to apheresis;
   * Venetoclax (BCL-2 inhibitor) within 4 d prior to apheresis;
   * Idelalisib (PI3Kδ kinase inhibitor) within 2 d prior to apheresis;
   * Lenalidomide within 1 d prior to apheresis;
   * Lymphocytotoxic chemotherapy within 2 weeks prior to apheresis - use in more than 3 half-lives prior to apheresis is eligible;
   * Non-lymphocytotoxic chemotherapy within 7 d prior to apheresis - use in more than 3 half-lives prior to apheresis is eligible;
   * Radiotherapy within 6 weeks prior to apheresis, including big bone marrow area (e.g., sternum or pelvis) - progressive disease at radiotherapy site, or PET positive lesion at other non-radiotherapy site is eligible; if there is existing PET positive lesion in other non-radiotherapy sites, then it is allowable to conduct radiotherapy at a single lesion within 2 weeks prior to apheresis.
4. Patients receiving chemotherapy within 2 weeks prior to CNCT19 Cell injection infusion, excluding the following conditions:

   * Pretreatment chemotherapy as specified by the protocol;
   * CNS lymphoma prophylaxis by intrathecal injection (it must be stopped within 1 week prior to infusion of CNCT19 Cell Injection).
5. Discontinuation of a systematic therapeutic hormone within 72 h prior to infusion of CNCT19 Cell Injection; however, use of the hormone in the physiological surrogate amount is eligible (e.g., Prednisone in a dose of <10 mg/d or equivalent).
6. Patients previously received CAR-T cell therapy.
7. Patients who have previously received allogeneic hematopoietic stem cell transplantation (allo-HSCT).
8. Patients with known active or uncontrolled synstemic autoimmune disease and under treatment.
9. Patients complying with any of hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive, hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive and HBV-DNA copies being more than the lower limit of detection, hepatitis C antibody (HCV-Ab) positive, anti-treponemia pallidum antibody (TP-Ab) positive, EBV-DNA, and CMV-DNA copies being more than the lower limit of detection.
10. Patients who received a major surgery within 4 weeks prior to screening, and are not eligible for enrollment as judged by the investigator.
11. Patients with concurrent active malignancy; those with a history of malignancy, cured for≥2 years, are eligible.
12. Patients complying any of the following conditions: Left ventricular ejection fraction (LVEF) ≤45% (ECHO); New York Heart Association (NYHA) Grade III or IV congestive heart failure; Uncontrolled hypertension (systolic blood pressures≥140mmHg and/or diastolic blood pressures ≥90 mmHg), pulmonary hypertension, or unstable angina pectoris; Myocardial infarction or bridging or stent procedure within 12 months prior to administration of the drug; Clinically significant valvular heart disease; Other heart diseases unsuitable for enrollment, as judged by the investigator.
13. Patients with lymphoma involved with atrium or ventricle.
14. Patients with clinical emergency (e.g., intestinal infarction or vascular compression) requiring treatment, due to existing lymphoma body obstruction or compression at screening.
15. Patients with active hemorrhage at screening.
16. Patients with deep vein thrombosis within 6 months prior to screening, or a history of pulmonary embolism.
17. Patients who are known with a history of hypersensitivity reaction to any ingredient used for the drug product in the trial.
18. Patients vaccinated with a live vaccine within 6 weeks prior to screening.
19. Patients with active infection at screening.
20. Patients with a life expectancy of less than 3 months.
21. Patients participating in any other interventional clinical study or receiving treatment of an active investigational drug within 3 half-lives prior to CNCT19 Cell Injection infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | At 3 months after infusion
  Efficacy of CNCT19 as measured by ORR at the 3 months after CNCT19 Cell Injection infusion, which includes CR and PR.

SECONDARY OUTCOMES:
CR rate at 3 months after CNCT19 infusion | 3 months
  Efficacy of CNCT19 as measured by CR during the 3 months after CNCT19 Cell Injection infusion.
ORR（CR+PR）/CR | 28 days
ORR（CR+PR）/CR | 6 months
Progression-free survival (PFS) | 24 months
  PFS means duration from the CNCT19 Cell Injection infusion to progression of lymphoma, or death for any reason.
Disease-free survival (DFS) | 24 months
  DFS means duration from the beginning of complete remission to relapse of disease, or death (for any reason).
Duration of Remission (DOR) | 24 months
  DOR means the duration from reaching the response (e.g., CR or PR) criteria of the therapy to the first, clearly defined progressive disease, or death for disease under investigation.
Best Overall Response (BOR) | 24 months
  The best overall response after CNCT19 infusion.
Overall Survival (OS) | 24months
  OS means duration from the CNCT19 Cell Injection infusion to death for any reason, or the last follow-up for survival.
Time to remission (TTR) | 24 months
  TTR means duration from the CNCT19 Cell Injection infusion to the first response (irrespective of PR or CR, which comes first).

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Weili Zhao, Dr., Principal Investigator — Ruijin Hospital
Locations (17):
- China (17):
  - Beijing Boren Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital of TMMU, Chongqing, Chongqing Municipality
  - Guangdong Provincial Peoples' Hospital, Guangzhou, Guangdong
  - SunYat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University school of Medicine, Hangzhou, Zhejiang